CLINICAL TRIAL: NCT00723346
Title: Administration of Allogenic of Red Blood Cells Loaded L Asparaginase in Acute Lymphoblastic Leukemia Relapse.
Brief Title: Administration of Allogenic Red Blood Cells Loaded L-asparaginase in Cases of Relapse of Acute Lymphoblastic Leukaemia
Acronym: GRASPALL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ERYtech Pharma (Industry)
Collaborators: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRASPALL 2005-01
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Relapse; Lymphoma lymphoblastic
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental)
  Interventions: Biological: GRASPA
- 2 (Experimental)
  Interventions: Biological: GRASPA
- 3 (Experimental)
  Interventions: Biological: GRASPA
- 4 (Active Comparator)
  Interventions: Drug: native L asparaginase

INTERVENTIONS:
Biological: GRASPA — 50 UI/Kg
  Arms: 1
Biological: GRASPA — 100 UI/Kg
  Arms: 2
Biological: GRASPA — 150 UI/Kg
  Arms: 3
Drug: native L asparaginase — 10000UI/m2, 14 infusions during 4 chemotherapy cycle
  Arms: 4

SUMMARY:
Primary objective :

* To explore the relation between 3 doses of GRASPA and duration of asparagine depletion (< 2µmol/l)

Secondary objective :

* Pharmacokinetic / Pharmacodynamic parameters
* toxicity
* Study duration : 2 years
* Study treatment : Red blood cells loaded with L asparaginase versus native L asparaginase
* Associated treatments : COPRALL chemotherapy
* Randomization : centralised randomisation on scratching list

ELIGIBILITY:
Inclusion Criteria:

* Subject between 1 and 55 year old
* Subject with acute lymphoblastic leukaemia or lymphoblastic lymphoma (excluded burkitt lymphoma) who have relapsed after first remission (medullary or SNC relapse)
* Or patient who still refractory to first line chemotherapy for an ALL
* Patient who gave written informed consent (2 parents for children)

Exclusion Criteria:

Ages: 1 Year to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2006-01; Primary Completion 2008-08 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Duration of plasmatic asparagin depletion (< 2µmol/l) | PK points

CONTACTS AND LOCATIONS:
Overall Officials: Yves Bertrand, MD PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hopital Debrousse, Lyon, France